CLINICAL TRIAL: NCT06913283
Title: Outcome of Pulpotomy Using Mineral Trioxide Aggregate and Biodentin in the Mature Permanent Teeth With Carious Exposure
Brief Title: Outcome of Pulpotomy With MTA and Biodentin in Permanent Teeth With Caries Exposure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Ambreen Mengal, Dentist AMengal, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Altamash IDM Ambreen
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — mineral trioxide aggregate; tricalcium silicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A Mineral trioxide aggregate pulpotomy (Active Comparator)
  Interventions: Procedure: Pulp Therapy with Mineral trioxide aggregate (MTA)
- Group B Biodentine pulpotomy (Active Comparator)
  Interventions: Procedure: Pulp Therapy with Biodentine

INTERVENTIONS:
Procedure: Pulp Therapy with Mineral trioxide aggregate (MTA) — MTA allowed to set for twenty four hours
  Arms: Group A Mineral trioxide aggregate pulpotomy
Procedure: Pulp Therapy with Biodentine — Biodentine is triturated before use
  Arms: Group B Biodentine pulpotomy

SUMMARY:
The success of pulpotomy treatment is affected by the type of biologically active material used.The effects of MTA and biodentine are compared in mature permanent teeth with caries exposure.It is expected that pulpotomy using biodentine will have a high success rate in caries exposed mature teeth compared to mineral trioxide aggregate.

ELIGIBILITY:
Inclusion Criteria:

* mature permanent teeth

Exclusion Criteria:

* Teeth with restorations

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated with MTA | 6 months
Number of Participants treated with Biodentine | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because it is mentioned in the patient consent form that details given by the patient and their identity will be kept confidential.